CLINICAL TRIAL: NCT05826639
Title: Risks, Safety, and Outcomes of Temperature-sensitive Endobiliary Radiofrequency Ablation in Patients With Malignant Biliary Obstructions
Brief Title: A Study of Endobiliary Radiofrequency Ablation in Malignant Biliary Obstructions
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Vinay Chandrasekhara, Principal Investigator, Mayo Clinic
Other Study IDs: 22-005206; NCI-2024-02188 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Biliary Stricture
Keywords: Bile duct obstruction; Biliary stent; Temperature-Sensitive Radiofrequency Ablation (RFA)
MeSH Terms: conditions — Cholestasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Temperature-sensitive RFA prior to biliary stenting: Data will be collected on subjects undergoing endoscopic retrograde cholangiopancreatography (ERCP) with temperature-sensitive RFA prior to biliary stenting for treatment of malignant biliary strictures as part of clinical care.
  Interventions: Procedure: Temperature-sensitive radiofrequency ablation
- Non-RFA biliary stenting for malignant biliary obstruction: Retrospective participants that have undergone non-RFA biliary stenting for malignant biliary obstruction from a historical cohort will serve as controls.
  Interventions: Other: No intervention

INTERVENTIONS:
Procedure: Temperature-sensitive radiofrequency ablation — Endobiliary radiofrequency ablation prior to ERCP-guided biliary stenting that utilizes a temperature-sensitive endobiliary RFA catheter
  Other Names: RFA
  Groups: Temperature-sensitive RFA prior to biliary stenting
Other: No intervention — No intervention
  Groups: Non-RFA biliary stenting for malignant biliary obstruction

SUMMARY:
The purpose of this study is to assess the impact of temperature-sensitive radiofrequency ablation (RFA) immediately before biliary stent placement on duration of biliary stent patency and re-intervention free survival. This is a research study meant to collect information to help other patients with malignant biliary strictures in the future.

ELIGIBILITY:
Inclusion Criteria:

* Malignant biliary stricture
* participants have or will have a biopsy-confirmed pancreaticobiliary or ampullary malignancy that have agreed to undergo radiofrequency ablation (RFA) with placement of biliary stents
* Patients with life expectancy greater than 3 months
* Able to provide consent

Exclusion Criteria:

* Patients who are pregnant
* Patients with cirrhosis
* Patients with significant liver metastasis >30% on radiologic imaging suggestive of poor liver function that will not improve despite endoscopic drainage.
* Patients who have undergone prior biliary decompression stents or percutaneous drainage that cannot be removed at time of ERCP and thus preclude effective RFA
* Patients with altered anatomy unable to undergo conventional ERCP (i.e., history of Roux-en-Y gastric bypass)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have or will have a biopsy-confirmed pancreaticobiliary or ampullary malignancy that have agreed to undergo radiofrequency ablation (RFA) with placement of biliary stents.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Stent patency | 6 months
  Duration of stent patency over the 6 month follow-up period
Re-intervention free survival | 6 months
  Duration of re-intervention free survival over the 6 month follow-up period
Mortality | 6 months
  Number of subject deaths following ERCP, over the 6-month follow-up period

SECONDARY OUTCOMES:
Adverse Events | 6 months
  Number of participants with treatment-related adverse events over the 6-month follow-up period
Time until first adverse event | 6 months
  Time (in days) from ERCP until first treatment-related adverse event, over the 6-month follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Chandrasekhara, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials